CLINICAL TRIAL: NCT06061302
Title: A Randomized Pilot Study of Yoga Intervention in Patients With Multiple Myeloma on Active Therapy
Brief Title: Multiple Myeloma Yoga Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003083
Record Dates: First submitted 2023-08-29; First posted 2023-09-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; yoga
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate yoga group (Experimental): 20 participants randomized to immediate yoga intervention group will participate together in a weekly 40-minute guided mindful yoga intervention for a total of 12 consecutive weeks. After each session, participants will be asked to complete the Edmonton Symptom Assessment System (ESAS-r) through MyDataHelps app. At the end of each session, participants will be asked additional questions via MyDataHelps such as completion of yoga session on-site or remotely, the length of time they participated in the session, any additional yoga sessions during the past week, and comments regarding the session/intervention. These participants will also complete health-related quality of life (HRQOL) assessment (EORTC QLQ-C30) at baseline, 6 weeks, and 12 weeks during active yoga intervention.
  Interventions: Other: Immediate yoga intervention
- Waitlist yoga group (delayed yoga intervention group) (Active Comparator): 20 participants randomized to this group will start the yoga intervention at week 13 and participate in 12 consecutive weeks of weekly 40 minute guided mindful yoga. Participants in this group will complete ESAS-r every 3 weeks and EORTC QLQ-C30 every 6 weeks for the first 12 weeks. These participants will also complete HRQOL assessment (EORTC QLQ-C30) at baseline, 6 weeks, and 12 weeks during active yoga intervention, weeks 13-24.
  Interventions: Other: Delayed yoga intervention

INTERVENTIONS:
Other: Immediate yoga intervention — Subjects will complete 12 consecutive weeks of weekly 40 minute guided mindful yoga weeks 1-12.
  Arms: Immediate yoga group
Other: Delayed yoga intervention — Subjects will complete 12 consecutive weeks of weekly 40 minute guided mindful yoga weeks 13-24.
  Arms: Waitlist yoga group (delayed yoga intervention group)

SUMMARY:
The purpose of this study is to evaluate the feasibility of implementing a weekly yoga intervention in patients with multiple myeloma on active therapy. This study aims to analyze the impact of yoga intervention on physical symptoms (e.g. pain, fatigue, sleep), psychological symptoms (e.g. anxiety, depression), and overall health-related quality of life (HRQOL) in multiple myeloma patients on active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any adult of age 18 and above
* Able to understand basic English
* Able to provide informed consent
* Diagnosis of multiple myeloma on active treatment as determined by investigators
* Good performance status as defined by European Cooperative Oncology Group score 0-1
* Able to utilize computer/laptop and smart phone
* Able and willing to travel to the yoga studio for weekly sessions
* Able to utilized a wearable device, such as Apple Watch or Fitbit (optional)

Exclusion Criteria:

* Poor performance status with European Cooperative Oncology Group score 2-4
* Actively participating in another clinical trial
* Poorly controlled mental health symptoms as determined by treating physician
* Reported fall or syncope in the last 2 months prior to enrollment
* Concurrent diagnosis of amyloidosis or other cancer requiring active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Compliance rate of weekly yoga intervention | 12 weeks
  Evaluate the feasibility of implementing a weekly 40-minute yoga intervention in patients with multiple myeloma on active treatment for 12 weeks by measuring compliance and overall completion rate of the program.
  Measurement: Compliance will be measured by overall percentage of patients completing 40 minutes of weekly yoga sessions in at least 8 out of 12 weeks of intervention. Completion rate will be measured by overall percentage of patients completing the 12 weeks of intervention without withdrawing or dropping out from the study.
  Hypothesis: Implementation of a weekly mindful yoga intervention will be feasible in multiple myeloma patients as demonstrated compliance of at least 70% patients completing 40 minutes of weekly yoga sessions in 8 out of 12 weeks of intervention.
Accrual rate of yoga intervention study | 12 weeks
  Evaluate the feasibility of implementing a weekly 40-minute yoga intervention in patients with multiple myeloma on active treatment for 12 weeks by measuring accrual rate.
  Measurement: Accrual rate will be measured by overall percentage of participants enrolled in the study at the end of 3-month accrual period compared to goal accrual of total 40 participants.
  Hypothesis: Implementation of a weekly yoga intervention will be feasible in multiple myeloma patients as demonstrated by accrual of 40 patients (100%) over 3 months.

SECONDARY OUTCOMES:
Short-term impact of yoga intervention on symptom burden | 12-weeks
  Evaluate the short-term impact of weekly yoga intervention in patients with multiple myeloma on active treatment on symptom burden by measuring Edmonton Symptom Assessment System (ESAS-r) after each session weekly.
  Measurement: Patient-reported scores will be measured after 40-minute yoga intervention each week using ESAS-r and they will be compared to baseline. Symptom assessment scale ranges from 0 (best) to 10 (worst).
  Hypothesis: Patients with multiple myeloma on active treatment will have statistically significant improvement in symptom burden compared to baseline after 40-minute yoga intervention each week.
Short-term impact of yoga intervention on health-related quality of life (HRQOL) | 12-weeks
  Evaluate the impact of a weekly 12-week yoga intervention program in patients with multiple myeloma on active treatment on health-related quality of life (HRQOL) over 12 weeks by measuring HRQOL questionnaire, European Organization For Research and Treatment Of Cancer-Core Quality of Life Questionnaire (EORTC QLQ-C30), responses at baseline, 6 and 12 weeks.
  Measurement: Overall health-related quality of life in participants will be measured at baseline, 6 and 12 weeks using EORTC QLQ-C30 assessment tool and scores will be compared to baseline. Scores range from 0 to 100 with higher numbers indicating higher function and quality of life. Subscale for symptom burden will indicate higher symptom burden with higher score values. Hypothesis: Patients with multiple myeloma on active treatment will have statistically significant improvement in HRQOL scores (measured by EORTC QLQ-C30) at 6 and 12 weeks compared to baseline and controls due to 12-week mindful yoga intervention.
Short-term impact of yoga intervention on total daily activity | 12-weeks
  Evaluate the impact of a 12-week mindful yoga intervention program in patients with multiple myeloma on active treatment on total daily activity measured by total daily steps using wearable device (FitBit).
  Measurement: Total daily steps will be measured in each participant using a wearable device (FitBit), and mean values from each week will be compared at baseline, 6 weeks, and 12 weeks.
  Hypothesis: Patients with multiple myeloma on active treatment undergoing yoga intervention will have increased total daily activity (daily steps) at 6 weeks and 12 weeks.
Short-term impact of yoga intervention on resting heart rate | 12-weeks
  Evaluate the impact of a 12-week mindful yoga intervention program in patients with multiple myeloma on active treatment on resting heart rate using wearable device (FitBit).
  Measurement: Resting heart rate will be measured in each participant using a wearable device (FitBit), and mean resting heart rate values from each week will be compared at baseline, 6 weeks, and 12 weeks.
  Hypothesis: Patients with multiple myeloma on active treatment undergoing yoga intervention will have decreased resting heart rate at 6 weeks and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Shaunak Pandya, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No